CLINICAL TRIAL: NCT02162550
Title: Effect of Bydureon on Carotid Atherosclerosis Progression in T2DM
Brief Title: Effect of Bydureon on Carotid Atherosclerosis Progression in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Phoenix VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter Reaven, Director, Diabetes Program, Phoenix VA Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1026
Record Dates: First submitted 2014-05-27; First posted 2014-06-12 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Cardiovascular Disease; Hyperglycemia; Carotid Plaque; Endothelial function; Incretins; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Hyperglycemia; Atherosclerosis | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bydureon (Experimental): injectable medication Bydureon
  Interventions: Drug: Bydureon
- Placebo (Placebo Comparator): a similar looking injectable
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bydureon — once weekly injection
  Other Names: long-acting exenatide
  Arms: Bydureon
Drug: placebo — once weekly injection
  Other Names: inactive agent
  Arms: Placebo

SUMMARY:
Investigators will be determining whether a once weekly injectable medication Bydureon versus placebo is able to reduce the development of atherosclerosis.

Investigators are testing the overall hypothesis that 18 months of Bydureon treatment will improve cardiovascular risk factors, endothelial function and retard carotid atherosclerosis plaque progression in type 2 diabetes mellitus (T2DM). Investigators anticipate these studies will provide novel information about the temporal relationship between Bydureon induced changes in risk factors, endothelial function and atherosclerosis progression.

DETAILED DESCRIPTION:
148 typical T2DM patients (ages 21-75) will participate in a rolling recruitment over approximately 2.25 years and be randomly allocated for 18 months to Bydureon (2 mg/week) or matching placebo subcutaneous injections 1x/week in a 2:1 ratio. Participants are expected to have a wide range of cardiovascular (CVD) risk and will therefore allow us to explore the importance of disease extent at baseline as a predictor of response. Blocked randomization will be used to ensure equal distribution of gender and CVD history. Carotid plaque MRI assessments will be performed at baseline, 9 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* males and females of any race and ethnicity with T2DM, HbA1c of ≥6.5% and ≤10.0% on diet only
* take stable doses of oral antihyperglycemic agents with or without long-acting insulin
* must have a regular primary care provider (PCP) that is amenable to patient study participation and will facilitate (blinded to the treatment) the research team's study protocol efforts

Exclusion Criteria:

* type 1 diabetes mellitus (T1DM)
* current or recent glucagon-like peptide 1 receptor (GLP-1R) agonist use
* contraindications to MRI (e.g., claustrophobia, ferromagnetic materials, body habitus inappropriate for MRI exam)
* screening carotid ultrasound plaque thickness of <0.75 mm, prior or anticipated carotid stenting or endarterectomy
* recent CVD (past 6 months) or other major illness or conditions affecting risk (e.g., pancreatitis, severe renal disease) or personal or family history of medullary thyroid carcinoma
* patients with Multiple Endocrine Neoplasia syndrome type 2
* serious hypersensitivity to exenatide or any product components
* severe gastrointestinal disease, or pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in carotid plaque volume | 18 months
  To determine the difference in change in carotid plaque volume, using 3 tesla (3T) MRI, between T2DM patients treated with Bydureon or placebo.

SECONDARY OUTCOMES:
Change in reactive hyperemic index | 18 months
  To determine the effects of long-term Bydureon therapy on vascular function as measured by the difference in fasting and post prandial reactive hyperemic index using peripheral artery tonometry.
Change in carotid plaque composition | 18 months
  To determine the difference in change in carotid plaque composition, using 3 tesla (3T) MRI, between T2DM patients treated with Bydureon or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Reaven, MD, Principal Investigator — Carl T. Hayden Medical Research Foundation
Locations (1):
- Phoenix VA Health Care System, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Subject to VA regulation.

REFERENCES:
- [Derived] Koska J, Migrino RQ, Chan KC, Cooper-Cox K, Reaven PD. The Effect of Exenatide Once Weekly on Carotid Atherosclerosis in Individuals With Type 2 Diabetes: An 18-Month Randomized Placebo-Controlled Study. Diabetes Care. 2021 Jun;44(6):1385-1392. doi: 10.2337/dc20-2014. Epub 2021 Jan 25. PMID 33495294